CLINICAL TRIAL: NCT07372209
Title: Study of Effects and Underlying Mechanisms of Analgesic Drugs on Inflammatory Pathways and Immune Function in Patients With Endometrial Cancer
Brief Title: Effects and Safety of Oliceridine in Anesthesia Induction:A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tangshan Maternal and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Yu Zhang, principle nvestigator, Tangshan Maternal and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-074-01
Record Dates: First submitted 2025-09-03; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Gynecological Laparoscopic Surgery; General Anesthetic; Intubation
MeSH Terms: interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sufentanil (Active Comparator): 0.5μg/kg of sufentanil was used for anesthesia induction
  Interventions: Drug: Sufentanil
- Oliceridine (Experimental): 0.13mg/kg oliceridine was used for anesthesia induction
  Interventions: Drug: Oliceridine

INTERVENTIONS:
Drug: Oliceridine — Oliceridine is diluted to a 1mg/kg injection solution
  Arms: Oliceridine
Drug: Sufentanil — sufentanil is diluted to a 5μg/ml injection solution
  Arms: sufentanil

SUMMARY:
to investigate whether oliceridine is safe and effective for induction of anesthesia by comparing henodynamic changes before and after endotracheal intubation with sufentanil

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years;
2. American Society of Anesthesiologists (ASA) physical status I-II;
3. Elective gynecologic laparoscopic surgery;
4. Expected operative time 60-180 minutes;

Exclusion Criteria:

1. Severe cardiovascular instability (e.g., acute decompensated heart failure, acute myocardial infarction, or life-threatening arrhythmia);
2. Uncontrolled hypertension;
3. Severe renal or hepatic dysfunction;
4. Severe mental disorder or psychiatric illness;
5. Known allergy or hypersensitivity to opioids;
6. History of alcohol abuse or opioid addiction;
7. Anticipated difficult airway;
8. Pregnancy or lactation;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
blood pressure | baseline, at the moment of intubation, right after intubation, 1 minute、3 minutes, and 5 minutes after intubation
heart beat | baseline, at the moment of intubation, right after intubation, 1 minute、3 minutes, and 5 minutes after intubation

SECONDARY OUTCOMES:
adverse reactions | from the administration of sufentanil or oliceridine until discharge from the post-anesthesia care unit (PACU)

CONTACTS AND LOCATIONS:
Locations (1):
- Tangshan Maternal and Child Health Hospital, Tangshan, Hebei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simons P, van der Schrier R, van Lemmen M, Jansen S, Kuijpers KWK, van Velzen M, Sarton E, Nicklas T, Michalsky C, Demitrack MA, Fossler M, Olofsen E, Niesters M, Dahan A. Respiratory Effects of Biased Ligand Oliceridine in Older Volunteers: A Pharmacokinetic-Pharmacodynamic Comparison with Morphine. Anesthesiology. 2023 Mar 1;138(3):249-263. doi: 10.1097/ALN.0000000000004473. PMID 36538359
- [Background] Paley EL. Phosphorylation of T antigen and p53 in carcinogen-treated SV40-transformed Chinese hamster cells. Carcinogenesis. 1996 May;17(5):939-45. doi: 10.1093/carcin/17.5.939. PMID 8640941
- [Background] Rahlfs S, Schirmer RH, Becker K. The thioredoxin system of Plasmodium falciparum and other parasites. Cell Mol Life Sci. 2002 Jun;59(6):1024-41. doi: 10.1007/s00018-002-8484-9. PMID 12169015
- [Background] Ma B, Li Y, Leng C, Ji A, Zhang N, Tao X, Cao Q, Wang S. A Comparative Evaluation of the Safety and Efficacy of Oliceridine and Sufentanil in Gastrointestinal Endoscopy: A Single-Center, Randomized Controlled Trial. Drug Des Devel Ther. 2025 Jun 17;19:5111-5121. doi: 10.2147/DDDT.S512529. eCollection 2025. PMID 40546662
- [Background] Iannuzzi E, Iannuzzi M, Cirillo V, Viola G, Parisi R, Cerulli A, Chiefari M. Peri-intubation cardiovascular response during low dose remifentanil or sufentanil administration in association with propofol TCI. A double blind comparison. Minerva Anestesiol. 2004 Mar;70(3):109-15. PMID 14997083
- [Background] Teong CY, Huang CC, Sun FJ. The Haemodynamic Response to Endotracheal Intubation at Different Time of Fentanyl Given During Induction: A Randomised Controlled Trial. Sci Rep. 2020 Jun 1;10(1):8829. doi: 10.1038/s41598-020-65711-9. PMID 32483139